CLINICAL TRIAL: NCT06829017
Title: Pilot Implementation and Evaluation of the Effectiveness of the Postoperative Hypothermia Management Care Bundle
Brief Title: Pilot Implementation of the Postoperative Hypothermia Management Care Bundle
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Ali Balkan, Research assistant, Hacettepe University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Record Dates: First submitted 2025-02-09; First posted 2025-02-17 (Actual); Last update posted 2025-07-25 (Actual); Status verified 2025-07

CONDITIONS: Postoperative Hypothermia
Keywords: postoperative hypothermia; care bundle; nursing; surgery; postoperative care

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- the pilot implementation and effectiveness of the postoperative hypothermia management care bundle (Other)
  Interventions: Other: Postoperative Hypothermia Management Care Bundle

INTERVENTIONS:
Other: Postoperative Hypothermia Management Care Bundle — The postoperative hypothermia care bundle consists of three main parameters, "Diagnose hypothermia", "Maintain/maintain normothermia" and "Monitor body temperature at regular intervals", and eight sub-parameters of these parameters. For this purpose, this study evaluates the pilot implementation and effectiveness of the postoperative hypothermia management care bundle developed within the scope of the research.

SUMMARY:
Inadvertent perioperative hypothermia (IPH) is a common complication in surgical patients, with incidence rates ranging between 50% and 90% in anaesthetised individuals. This study aims to pilot and evaluate the effectiveness of a Postoperative Hypothermia Management Care Bundle developed based on standardised, evidence-based practices.

The study will be conducted using a mixed-methods design in two phases.

In the first phase, the care bundle will be piloted over six months in the Cardiovascular Surgery Intensive Care Unit.

In the second phase, the bundle's effectiveness will be assessed using both quantitative and qualitative data.

The study population includes nurses working in the relevant intensive care unit who meet inclusion criteria and volunteer to participate.

Data collection tools include:

Nurse Descriptive Information Form

Postoperative Hypothermia Management Care Bundle Checklist

Care Bundle Compliance Assessment Form

Semi-structured Nurse Interview Questionnaire (qualitative)

Patient Postoperative Hypothermia Follow-up Form

Quantitative data will be analysed using descriptive statistics. Compliance with the care bundle will be calculated as the ratio of patients who received all care bundle parameters to those who should have received them. A compliance rate below 95% will be considered unsuccessful. Qualitative data will be analysed using Colaizzi's seven-step phenomenological method.

DETAILED DESCRIPTION:
Background and Rationale

Inadvertent perioperative hypothermia (IPH) is one of the most common perioperative problems in surgical patients. In the literature, IPH rates in anesthetized patients are reported between 50-90%. Guidelines for preventing and managing IPH in surgical patients have been developed. Although there are clinical practice guidelines for the management of IPH, the incidence of IPH in surgical patients is still high. Reducing the incidence of IPH in surgical patients depends on good management of hypothermia in the perioperative process, and nurses have important responsibilities at every stage of the perioperative process in the management of IPH. Nurses, who play a key role in the multidisciplinary team in the management of IPH, still experience some problems in the management of hypothermia. Good management of IPH, which is a preventable problem in the surgical process, may be possible with evidence-based standardization of practices in the perioperative process and systematic implementation of these practices.

Care Bundles for Hypothermia Management

In recent years, Care Bundles (CB) have been used to standardize nursing practices based on evidence and to improve the quality of care. CB is defined as a set of evidence-based practices used to standardize care and treatment. CBs are reported to have many benefits such as providing easy management of conditions requiring special care, reducing complications, increasing communication within the team, improving the quality of care, and providing supervision. In addition, it has been reported that the use of CB increases the satisfaction of patients and nurses and job satisfaction of nurses, reduces unnecessary applications in nursing care, and improves negative patient outcomes that may result from inadequate care. In the literature, there is a CB developed for the management of perioperative hypothermia. The perioperative thermal CB developed by Duff et al. (2018) includes three elements: risk assessment, body temperature monitoring, and active warming. The three elements in this CB are recommendations for preoperative, intraoperative, and postoperative processes, and it is evident that the majority of the applications are for the intraoperative phase. In the study, it was found that compliance with the CB, especially the practices in the intraoperative process, was low. It is thought that the development and use of a CB specific to each stage of the perioperative process in the management of IPH will increase the applicability of the CB and compliance with the bundle. In the literature, there is no CB developed for the management of hypothermia in the postoperative period. Therefore, a CB specific to the postoperative process was developed to standardize nursing care for hypothermia in surgical patients, improve patient outcomes, and increase the quality of care. This CB was prepared in line with the approaches recommended by the Institute for Healthcare Improvement (IHI) for the management of postoperative hypothermia.

Study Objectives This study evaluates the pilot implementation and effectiveness of the postoperative hypothermia management CB developed within the scope of the research.

Study Design and Setting This study was planned as mixed-method research in which qualitative and quantitative research methods were used together. The study is planned to be conducted in the Cardiovascular Surgery Intensive Care Unit of Hacettepe University Adult Hospital between 15 August 2025 and 31 March 2026 following the approval of the ethics committee.

Participants and Eligibility Criteria Participants include nurses working in the Cardiovascular Surgery Intensive Care Unit and patients hospitalized there. Inclusion criteria for nurses include at least 6 months working experience in the unit and voluntary participation. Patients must be 18 years or older, within the first 24 hours of postoperative follow-up, and must consent to participate.

Intervention: Postoperative Hypothermia Care Bundle The postoperative hypothermia CB consists of three main parameters: 'Diagnose hypothermia', 'Maintain/maintain normothermia', and 'Monitor body temperature at regular intervals', and eight sub-parameters. The CB was developed using literature review, expert consultation through Delphi method, and finalized after two rounds with 11 experts.

Data Collection Tools

1. Nurse Descriptive Information Form
2. Postoperative Hypothermia Management Care Bundle Checklist
3. Compliance Assessment Form
4. Semi-structured Questionnaire for Nurses
5. Patient Postoperative Hypothermia Follow-up Form

Procedure The study will be conducted in two phases: (1) pilot implementation of the CB and (2) evaluation of its effectiveness. Nurses will be trained and asked to use the CB checklist during their shifts for six months. Researchers will assess compliance and conduct qualitative interviews to evaluate nurse experiences. Data on hypothermia incidence and normothermia recovery time will also be collected.

Data Analysis Quantitative data will be analyzed using SPSS 23.0; descriptive statistics will be presented as means, standard deviations, medians, and percentages. Qualitative data will be analyzed using Colaizzi's seven-step phenomenological method. Compliance with the CB will be calculated and compared against a 95% threshold to assess success.

ELIGIBILITY:
Inclusion Criteria:

For Nurses

* Working as a nurse in Cardiovascular Surgery Intensive Care Unit for at least 6 months
* Volunteering to participate in the study

For patients to be cared for during the pilot implementation of the care bundle:

* 18 years of age or older
* Being in the first 24 hours of postoperative follow-up in the Cardiovascular Surgery Intensive Care Unit
* He/she or his/her legal representative has given consent to participate in the study

Exclusion Criteria:

For nurses

* Leaving the Cardiovascular Surgery Intensive Care Unit before the completion of the study period
* Unwillingness to continue working

For patients to be cared for during the piloting of the care package:

- Emergency surgical operations, patients with abnormal thermoregulation such as malignant hyperthermia and neuroleptic malignant syndrome and patients with ASA IV-V

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-15 (Estimated); Primary Completion 2026-02-15 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Care bundles compliance assessment form for postoperative hypothermia management | 15 August 2025-28 February 2026
  This form was developed by the researchers to evaluate the nurses' application of the care bundle to the patients. The boxes 'applied', 'not applied' if not applied, and 'not filled' if the control form is not marked will be ticked on the compliance assessment form in which the care bundle parameters are applied. Within the scope of this form, the compliance rate of the care bundle will be calculated. The rate found with this calculation will show the success of compliance with the maintenance bundle. In the calculation, the compliance rate will be calculated by dividing the number of patients to whom all parameters of the care bundle are fully implemented within the scope of the research by the number of patients to whom the care bundle parameters should be implemented. In this calculation, if the compliance rate is below 95%, it means that compliance with the care bundle is unsuccessful.

CONTACTS AND LOCATIONS:
Overall Officials: Zeliha OZDEMIR KOKEN, ASSOCIATE PROFESSOR, Study Director — Hacettepe University Faculty of Nursing; Mustafa YILMAZ, PROFESSOR, Study Chair — Hacettepe University Medicine Faculty
Locations (1):
- Hacettepe University adult hospital, Ankara, ABD Veya Kanada'daysanız Lütfen Seçin..., Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided